CLINICAL TRIAL: NCT03488940
Title: Effect of Different Feeding Method on Gastrointestinal Function of Septic Patients (DFM-GF Trial)
Acronym: DFM-GF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects were enrolled in other studies about sepsis
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Guang Yang, Director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFM-GF Trial
Record Dates: First submitted 2017-05-25; First posted 2018-04-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Sepsis; Intestinal Dysfunction
Keywords: Sepsis; intestinal dysfunction; enteral feeding
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 24-hours group (Active Comparator): The septic patients randomized to 24-hours group will be received enteral nutrition preparation by 24 hours of continuously pumping through stomach tube every day.
  Feeding will be started within 24 hours in admission of ICU. The time of therapy is 7 days.
  Interventions: Device: 24-hours group
- 16-hours group (Experimental): The septic patients randomized to 16-hours group will be received enteral nutrition preparation by 16 hours of continuously pumping through stomach tube every day.
  Feeding will be started within 24 hours in admission of ICU. The time of therapy is 7 days.
  Interventions: Device: 16-hours group
- intermittent group (Experimental): The septic patients randomized to intermittent group will be received enteral nutrition preparations by four meals every day(08:00,12:00 18:00,22:00), each meal are pumped within 60mins through stomach tube.
  Feeding will be started within 24 hours in admission of ICU. The time of therapy is 7 days.
  Interventions: Device: intermittent group

INTERVENTIONS:
Device: 24-hours group — Daily amount of feeding were continuously pumped for 24 hours. Enteral nutrition preparations pumping scheme: the initial pumping speed is 40ml/h, and gastric residual volumes(GRV) is checked every 4 hours. If it can be tolerated, the velocity of the pumping can be increased by half of the original speed.If it is not tolerable, the speed of the pumping is reduced by half on the original speed.
  GRV<200 mL were considered markers of good tolerance. Feeding intolerance was defined as GRV>200 mL.
  Enteral nutrition preparation are Enteral Nutritional Suspension(TPF-FOS) which were producted by ABBOTT LABORATORIES B.V.. The feeding pump are Infusion pump P-600 which were producted by Atom Medical Corporation.
  Other Names: Continuously-feeding pumped in 24 hours group
  Arms: 24-hours group
Device: 16-hours group — Daily amount of feeding were continuously pumped for 24 hours.Enteral nutrition preparations pumping scheme: the initial pumping speed is 40ml/h, and gastric residual volumes is checked every 4 hours. If it can be tolerated, the velocity of the pumping can be increased by half of the original speed.If it is not tolerable, the speed of the pumping is reduced by half on the original speed.
  GRV<200 mL were considered markers of good tolerance. Feeding intolerance was defined as GRV>200 mL.
  Enteral nutrition preparation are Enteral Nutritional Suspension(TPF-FOS) which were producted by ABBOTT LABORATORIES B.V.. The feeding pump are Infusion pump P-600 which were producted by Atom Medical Corporation.
  Other Names: Continuously-feeding pumped in 16 hours group
  Arms: 16-hours group
Device: intermittent group — Daily amount of feeding were divided into four meals, each meal are pumped within 60mins through stomach tube.
  Enteral nutrition preparations pumping scheme: the initial pumping speed is 200ml/h, and gastric residual volumes is checked before each intermittent feeding. If it can be tolerated, the velocity of the pumping can be increased by half of the original speed.If it is not tolerable, the speed of the pumping is reduced by half on the original speed.
  GRV<200 mL were considered markers of good tolerance. Feeding intolerance was defined as GRV>200 mL.
  Enteral nutrition preparation are Enteral Nutritional Suspension(TPF-FOS) which were producted by ABBOTT LABORATORIES B.V.. The feeding pump are Infusion pump P-600 which were producted by Atom Medical Corporation.
  Other Names: intermittent-feeding pumped group
  Arms: intermittent group

SUMMARY:
The intestine is the most vulnerable target organ in septic patients and is the first to be damaged organ in multiple organ dysfunction syndrome(MODS). Therefore, improving intestinal motility and mucosal barrier function is critical to the treatment of sepsis. Many studies have shown that, early enteral nutrition(EN) in patients with sepsis helps prevent and treat intestinal dysfunction, reducing ICU mortality and length of stay in ICU. However, there is little research on feeding methods. In this study we will compare the outcomes of different feeding methods: continuously-pumped in 24 hours, continuously-pumped in 16 hours and intermittently-pumped through the stomach tube. The aim of this study is to investigate the effects of different feeding methods on intestinal function in septic patients.

DETAILED DESCRIPTION:
Sepsis is the major cause of death in intensive care unit(ICU). According to the latest literature statistics in 2012, the mortality of sepsis was growing at 2% a year in the United States, and the average hospitalization costs of septic patients was more than $20000. Sepsis has become one of the big challenges to doctors in ICU all over the world. Previous studies found that intestinal dysfunction may be the main promoter and stimulating factor of systemic inflammatory response syndrome(SIRS), which plays an important role of in the development of sepsis to multiple organ dysfunction syndrome(MODS). But at present there is no effective treatment of intestinal dysfunction. Nutrient intake is considered part of the resuscitation of critical patients. Enteral feedings are considered standard treatment of the critically ill patients. A number of study have found enteral feedings could cure intestine dysfunction through improving circulation perfusion and oxygen delivery, maintaining intestinal mucosal barrier, reconstructing intestinal continuity and adjusting internal environment. Recent clinical researches and guidelines pointed out the importance of early enteral nutrition. However, guidelines made no mention of how to carry on the feeding method in severe patients, and related research is few.The current research mostly thinks, enteral nutrition preparations continuously pumped by stomach tube is a more accepted way.The researches cited by the guideline showed that the continuous feeding was better than that of intermittent feeding. But 24 hours of continuous pumping nutrition preparation will not only cause continuous stimulation to the intestinal mucosa, but also lead to gastrointestinal tract have not rest time. Some previous studies found intermittent feedings were better than continuous feedings to critical patients. So，was intermittent feeding really better? Therefore this research will compare the results of different feeding methods of EN: continuously-pumped in 24 hours, continuously-pumped in 16 hours and intermittently-pumped through the stomach tube. Then observe the effects of different feeding methods on intestinal function in septic patients so as to offer a more suitable EN feeding method for septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Septic patients in Department of Critical Care Medicine, Guangdong Provincial Hospital of Chinese Medicine;
2. APACHE-Ⅱ score greater than 15 points;
3. Signing the informed consent.

Exclusion Criteria:

1. Fasting patients in the clinical, such as digestive tract perforation, bleeding or postoperative patients with gastrointestinal tract;
2. Allergic to enteral nutrition preparations;
3. Early stage of sepsis (within a week) patients with hemodynamic instability;
4. Don't want to attend the test or not with the healer.

Fall Off Criteria:

1.Time is less than 7 days in hospital.

Suspension or Termination Criteria:

1.The patients can't tolerate enteral nutrition preparations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
The mean time(hours) that reach to the caloric goal in every group. | First 7 days after intervention
  Caloric goals using 25 kcal/kg (ideal body weight) for caloric need calculated by a single nutritionist.

SECONDARY OUTCOMES:
The rate of onset of Gastric residual (%) | First 7 days after intervention
  The definition of gastric residual is that gastric residual volume more than 500 ml. Comparison of rate of gastric residual among three groups.
Abdominal pressure (mmHg) | baseline and 7 days
  Abdominal pressure measurement: through the bladder indirect pressure measurement method, first taking the supine position, emptying the bladder urine, secondly pouring 50ml saline into the balloon catheter, to the pubic symphysis as the base point, keeping the piezometric tube be perpendicular to the ground, then abdominal pressure can be obtained indirectly.
Motilin (MTL) (pg/ml) | baseline and 7 days
  the level of plasma MTL
the rate of new onset pneumonia (%) | First 7 days after intervention
  Diagnosis of onset pneumonia is defined as two of the following clinical criteria were required. Fever (>38.3℃) or hypothermia (≤36.0℃), leukocytosis (>10×10E9 cells/liter) or leukopenia (≤4×10E9 cells/liter), purulent tracheal aspirate or sputum. The rate of onset pneumonia be counted in each group.
The rate(%) of people whom can reaching the caloric goal. | First 7 days after intervention
  Caloric goals using 25 kcal/kg (ideal body weight) for caloric need calculated by a single nutritionist.

OTHER OUTCOMES:
length of ICU stay (in days) | up to 12 weeks
  length of ICU stay (in days)
ICU mortality rate (%) | 28 days after intervention
  ICU mortality rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Study Chair — 2nd Affiliated Hospital of Guangzhou University of Chinese Medicine
Locations (1):
- 2nd Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Sharing data can be used by retrospective analysis and systematic review about intestinal dysfunction or septic patients starting in January 2022.The data including age, gender, damaged organs, basic disease, APACHE-II score, target calories, the time to reach target calories, gastric residual volume, abdominal pressure (cmH2O), level of plasma motilin(pg/ml), level of plasma intestinal fatty acid binding protein, intestinal dysfunction score, new onset pneumonia, duration of ICU and prognosis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Three years after the end of the study (starting in January 2022)
Access Criteria: Sharing data can be used by retrospective analysis, mechanism research and systematic reviews about intestinal dysfunction or septic patients. The researchers should be clinicians or medical researchers of respirology, intensive care medicine or gastroenterology.

REFERENCES:
- [Background] Lagu T, Rothberg MB, Shieh MS, Pekow PS, Steingrub JS, Lindenauer PK. Hospitalizations, costs, and outcomes of severe sepsis in the United States 2003 to 2007. Crit Care Med. 2012 Mar;40(3):754-61. doi: 10.1097/CCM.0b013e318232db65. PMID 21963582
- [Background] Nieuwenhuijzen GA, Deitch EA, Goris RJ. The relationship between gut-derived bacteria and the development of the multiple organ dysfunction syndrome. J Anat. 1996 Dec;189 ( Pt 3)(Pt 3):537-48. PMID 8982828
- [Background] Pastores SM, Katz DP, Kvetan V. Splanchnic ischemia and gut mucosal injury in sepsis and the multiple organ dysfunction syndrome. Am J Gastroenterol. 1996 Sep;91(9):1697-710. PMID 8792684